CLINICAL TRIAL: NCT06780865
Title: Protection of Renal Function by Antihypertensive Treatment in Patients with Chronic Kidney Disease and Isolated Nighttime Hypertension
Brief Title: Protecting Renal Function in Chronic Kidney Disease Patients with Isolated Nighttime Hypertension
Acronym: PRECISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Hypertension (Other)
Responsible Party: Principal Investigator, Yan Li, Professor, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRECISE Trial
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease(CKD); Nocturnal Hypertension
Keywords: chronic kidney disease; isolated nocturnal hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — arotinolol; Amlodipine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-hypertensive treatment group (Experimental): The patients will be treated with Arotinolol and/or Amlodipine and/or Clonidine.
  Interventions: Drug: Antihypertensive treatment with Arotinolol or Amlodipine or Clonidine
- Control group (Placebo Comparator): Placebo was used in the control group.
  Interventions: Drug: Placebo-controlled group

INTERVENTIONS:
Drug: Antihypertensive treatment with Arotinolol or Amlodipine or Clonidine — Participants will receive Almar 10 mg orally once daily between 8:00 PM and midnight. At the subsequent visit, if nocturnal blood pressure remains above the target of <120/70 mmHg, Amlodipine Besylate will be added at a dose of 2.5 mg to 5 mg orally once daily. Should nocturnal blood pressure still not achieve the target at the following visit, Clonidine Hydrochloride 75 µg will be added to the regimen. The target for nocturnal blood pressure control is set at <120/70 mmHg. For participants whose clinic blood pressure exceeds 140/90 mmHg, an unscheduled visit will be arranged within one month. If elevated clinic blood pressure persists during this visit, a 24-hour Ambulatory Blood Pressure Monitoring (ABPM) will be conducted. If the ABPM results indicate daytime blood pressure ≥135/85 mmHg, open-label add-on antihypertensive therapy will be initiated, prioritizing the use of antihypertensive medications outside of the study drugs to achieve blood pressure control.
  Arms: Anti-hypertensive treatment group
Drug: Placebo-controlled group — Participants are treated with corresponding placebo
  Arms: Control group

SUMMARY:
Hypertension guidelines recommend the application of ambulatory blood pressure monitoring in the diagnosis and treatment of patients with hypertension. Subtypes of hypertension such as nocturnal hypertension can be found through ambulatory blood pressure monitoring. Previous studies have reported that the prevalence of nocturnal hypertension, even isolated nocturnal hypertension, is higher in patients with chronic kidney disease, and it is associated with adverse events such as cardiovascular events and progression of renal dysfunction. However, the benefit of controlling nocturnal hypertension in patients with chronic kidney disease is unclear. In this study, a total of 200 patients with chronic kidney disease and isolated nocturnal hypertension will be enrolled. Patients will be randomly divided into two treatment groups: the active antihypertensive treatment group and the placebo treatment group (1:1). The antihypertensive treatment group will be treated with arotinolol or amlodipine and clonidine to control nocturnal blood pressure, while the control group will be treated with the corresponding placebos. Randomized patients will be followed up for 2 years to evaluate the effect of controlling isolated nocturnal hypertension on the progression of chronic kidney disease in terms of EPI-estimated glomerular filtration rate (eGFR) decline and change in proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older. All genders are eligible;
* Confirmed diagnosis of Chronic Kidney Disease (CKD) according to KDIGO. guidelines;
* UACR < 30 mg/g (3.4 mg/mmol) and eGFR between 20-44 mL/min/1.73 m²; or UACR between 30-300 mg/g (3.4-33.9 mg/mmol) and eGFR between 20-59 mL/min/1.73 m²; or UACR between 300-5000 mg/g (33.9-565 mg/mmol) and eGFR > 20 mL/min/1.73 m² (CKD-EPI equation).
* Office blood pressure measurements below 140/90 mmHg at both screening visits;
* Daytime ambulatory blood pressure < 135/85 mmHg and nighttime systolic blood pressure ≥ 120 mmHg or diastolic blood pressure ≥ 70 mmHg;
* No use of corticosteroids, immunosuppressants, or biologic agents for at least one month prior to enrollment;

Exclusion Criteria:

* Presence of acute kidney injury or acute renal failure;
* History of kidney transplantation;
* Presence of severe arrhythmias, including severe atrial fibrillation, atrioventricular (AV) block, sinoatrial (SA) block, sinus bradycardia, malignant AV node reentrant tachycardia syndrome;
* Secondary hypertension related to suspected or confirmed renal artery stenosis or adrenal gland disorders;
* Poor glycemic control (HbA1c > 12%);
* Orthostatic hypotension (a decrease in blood pressure of >20/10 mmHg within 3 minutes of standing from a sitting position);
* Women who are pregnant or breastfeeding at the time of enrollment, or not employing contraception of reproductive age;
* NYHA (New York Heart Association) Class III-IV congestive heart failure at the time of enrollment;
* History of myocardial infarction, unstable angina, acute heart failure, stroke, transient ischemic attack (TIA), or cerebral hemorrhage within the 12 weeks prior to enrollment;
* Underwent coronary revascularization (Percutaneous Coronary Intervention [PCI] or Coronary Artery Bypass Grafting [CABG]), or valve repair/replacement within the 12 weeks prior to enrollment, or planned to undergo any of the aforementioned surgical procedures after randomization;
* Any other serious diseases outside the renal and cardiovascular domains, including but not limited to malignancies, with an expected survival of less than 2 years based on the investigator's clinical judgment;
* Presence of active malignancy requiring pharmacological treatment;
* AST (Aspartate Aminotransferase) or ALT (Alanine Aminotransferase) levels >3 times the upper limit of normal (ULN);
* Total bilirubin >2 times ULN. Patients with Gilbert's syndrome who exhibit isolated bilirubin elevation do not need to be excluded;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in renal function from baseline after 2 year of treatment as assessed by EPI-estimated glomerular filtration rate (eGFR) | 2 years

SECONDARY OUTCOMES:
Change in renal function from baseline after 1 year of treatment as assessed by EPI-estimated glomerular filtration rate (eGFR) | 1 year
Change in urine protein from baseline after 1 and 2 years of treatment as assessed by urinary albumin-to-creatinine ratio(UACR) | 1 and 2 years
50% decrease of albumin-to-creatinine ratio (UACR) from baseline after 1 and 2 years of treatment | 1 and 2 years
Incidence of kidney composite endpoint including end-stage renal disease (ESRD), kidney replacement therapy, or sustained EPI-estimated glomerular filtration rate (eGFR) decline ≥ 40%. | 1 and 2 years
Incidence of sustained EPI-estimated glomerular filtration rate (eGFR) < 15 ml/min/1.73 m² | 1 and 2 years
Incidence of cardiovascular endpoints including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, or heart failure hospitalization | 1 and 2 years
Changes in cardiac injury after 1 and 2 years of treatment from baseline as assessed by left ventricular mass index or E/E' or cardiac troponin | 1 and 2 years
Changes in pulse wave velocity (PWV) after 1 and 2 years of treatment from baseline | 1 and 2 years
Incidence of mortality including all-cause, cardiovascular-related, and renal-related. | 1 and 2 years
Changes in office and ambulatory blood pressure levels after 1 and 2 years of treatment from baseline | 1 and 2 years
Hypotension-related adverse events | 1 and 2 years
  dizziness, falls, office blood pressure below 90/60 mmHg, orthostatic hypotension (blood pressure drop exceeding 20/10 mmHg within 3 minutes of standing compared to sitting), and acute kidney injury [serum creatinine increase ≥0.3 mg/dl (≥26.5 μmol/L) within 48 hours; or serum creatinine rising to ≥1.5 times baseline value within 7 days; or urine output <0.5 mL/(kg·h) for ≥ 6 hours].

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Palevsky PM, Liu KD, Brophy PD, Chawla LS, Parikh CR, Thakar CV, Tolwani AJ, Waikar SS, Weisbord SD. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for acute kidney injury. Am J Kidney Dis. 2013 May;61(5):649-72. doi: 10.1053/j.ajkd.2013.02.349. Epub 2013 Mar 15. PMID 23499048
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Buckalew VM Jr, Berg RL, Wang SR, Porush JG, Rauch S, Schulman G. Prevalence of hypertension in 1,795 subjects with chronic renal disease: the modification of diet in renal disease study baseline cohort. Modification of Diet in Renal Disease Study Group. Am J Kidney Dis. 1996 Dec;28(6):811-21. doi: 10.1016/s0272-6386(96)90380-7. PMID 8957032
- [Background] Chen N, Wang W, Huang Y, Shen P, Pei D, Yu H, Shi H, Zhang Q, Xu J, Lv Y, Fan Q. Community-based study on CKD subjects and the associated risk factors. Nephrol Dial Transplant. 2009 Jul;24(7):2117-23. doi: 10.1093/ndt/gfn767. Epub 2009 Feb 4. PMID 19193736
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068